CLINICAL TRIAL: NCT03841929
Title: Multimodal Monitoring of Hemodynamics in Extremely Low Birth Weight Preterm Infant in a Canadian Tertiary Level Unit- Non-Blinded Randomized Control Trial
Brief Title: Multimodal Monitoring of Hemodynamics in Extremely Low Birth Weight Preterm Infant in a Canadian Tertiary Level Unit
Acronym: MUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Kumar Kumaran, Clinical Associate Professor, University of Alberta,, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00084238
Record Dates: First submitted 2019-02-05; First posted 2019-02-15 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hemodynamic Instability
Keywords: Multimodal hemodynamic assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): ELGANs recruited to the study group in addition to standard of care will have continuous cerebral NIRS monitoring for the initial 72 hours and TNE studies at definitive time frames and a hemodynamic report will be provided to the clinical team using the results of the multimodal monitoring and clinical data. The report will be a description of the hemodynamic status without any suggestions for management.
  Interventions: Other: Hemodynamic report
- Standard Arm (No Intervention): ELGANs recruited into Standard arm will have the standard monitoring including cardiorespiratory monitoring. The invasive blood pressure monitoring, NIRS and TNE monitoring as per the clinical team's discretion - consistent with the current standard of care. No hemodynamic report will be provided routinely.

INTERVENTIONS:
Other: Hemodynamic report — The multimodal data comprising the clinical, biochemical, NIRS data and TNE where available will be used by the study team in such cases to reach a description of the hemodynamic status of the study infant and will be provided to the Clinical team.
  Arms: Study Arm

SUMMARY:
Low blood pressure is a common problem in the premature newborn and can affect over 30% of all Extremely Low Gestational Age Neonates (ELGAN) babies delivered less than 28 weeks completed. Neonatal clinicians assess the hemodynamic status of the infant using clinical signs and physiological parameters including heart rate, blood pressure, capillary refill time, urine output and laboratory parameters (base deficit and lactate). While urine output and laboratory parameters do not provide real-time assessment of the hemodynamic status, heart rate and capillary refill time could be non-specific, inaccurate and observer-dependent, respectively. Blood pressure (BP) continues to be used as a common physiological marker for cardiovascular state in neonates.However, there is increasing amount of evidence that monitoring blood pressure alone is not enough to ensure adequate systemic and cerebral perfusion and oxygenation. Indeed, preterm babies may have "low blood pressure" triggering pharmacological treatment while still maintaining adequate systemic flow- especially cerebral and other organ perfusion as shown by other noninvasive measures like targeted neonatal echocardiography (TNE) and near infrared spectroscopy (NIRS).

Using mean BP alone as the indication of treatment of neonatal cardiovascular compromise without taking into consideration the status of tissue perfusion may lead to unnecessary exposure of neonates to vasoactive medication. This medication can be potentially harmful to these extremely vulnerable patients. Analysis of a large neonatal database has demonstrated that treatment of hypotension was associated with an increase in serious brain injury. This held true even after the blood pressure was included in the regression mode, suggesting that it is treatment of hypotension, rather than the presence of hypotension which is harmful. The common interventions, fluid boluses followed by inotropes, could as well be harmful. Observational data has shown an association of fluid boluses with intracranial bleeding and in animal models intraventricular haemorrhage after hypotension can be induced by rapid volume infusion. Fluctuations in blood pressure when inotropes are introduced are well known and could also trigger haemorrhage.

Current standard approaches to evaluation and treatment of transitional circulatory problems in the preterm infant may be harmful. Therefore it is essential that these approaches are adequately investigated. This research study is trying to find out if having a detailed hemodynamic understanding using a multimodal assessment consisting of Targeted Neonatal Echocardiogram, Cerebral NIRS and clinical-biochemical data, will result in less inotrope use in ELGAN population during the first 72hours of transitional period.

DETAILED DESCRIPTION:
Background:

Neonatal transition from the intra-uterine to extra-uterine environment is a complex, multi-organ process. The heart of a term neonate is anatomically and functionally mature to make the transition. However, the feto-neonatal transition of Extremely Low Gestational Age Neonates (ELGAN) may have significant challenges in the context of the physiologically "less than adequate" myocardial function and a delicate balance between pulmonary and systemic blood flow. Further, the brain and cerebrovascular state of ELGAN are particularly vulnerable to the effects of an unbalanced transition. Despite advances in neonatal intensive care that have contributed to a decline in mortality and morbidity, preterm birth remains a major cause of mortality and long term neurological sequelae. Brain injury in preterm infants is often caused by disturbances in cerebral blood flow (CBF) and oxygenation that happen early in the transition when the majority of intraventricular bleeds and parenchymal infarcts occur. Therefore, it is important to evaluate the systemic and regional hemodynamic state of ELGAN in order to facilitate the neonatal transition.

Neonatal clinicians assess the hemodynamic status of the infant using clinical signs and physiological parameters including heart rate, blood pressure, capillary refill time, urine output and laboratory parameters (base deficit and lactate). While urine output and laboratory parameters do not provide real-time assessment of the hemodynamic status, heart rate and capillary refill time could be non-specific, inaccurate and observer-dependent, respectively. Blood pressure continues to be used as a common physiological marker for cardiovascular state in neonates. However, there is increasing amount of evidence that monitoring blood pressure alone is not enough to ensure adequate systemic and cerebral perfusion and oxygenation. Indeed, preterm babies may have "low blood pressure" triggering pharmacological treatment while still maintaining adequate systemic flow- especially cerebral and other organ perfusion as shown by other noninvasive measures like targeted neonatal echocardiography (TNE) and near infrared spectroscopy (NIRS). Interestingly, studies have demonstrated that independent of early blood pressure changes, anti-hypotensive therapy exposure in ELGAN was associated with an increased risk of death/NIDD at 18-22 months' corrected age even after controlling for risk factors known to affect survival and neurodevelopment.

The use of targeted neonatal echocardiography (TNE) by neonatal clinicians to evaluate cardiovascular state in neonates is common in many tertiary neonatal intensive care units. When used in combination with clinical findings, neonatal echocardiography may be an invaluable tool for the identification of hemodynamic compromise, guiding therapeutic intervention, and monitoring treatment response. There are an increasing number of prospective studies that highlight the potential merits of TNE in identification of cardiovascular compromise and guiding neonatal cardiovascular care. In addition, it has been shown that the use of early echocardiography to provide targeted PDA treatment may result in a reduction of severe intraventricular hemorrhage and pulmonary hemorrhages. The role of TNE to study organ blood flow including cerebral, renal and the gut is largely limited.

Near-infrared spectroscopy (NIRS) is a technique that can be used to monitor regional cerebral oxygen saturation (rScO2), being both a measure of cerebral oxygenation as well as a surrogate of cerebral blood flow. NIRS monitoring can be applied for prolonged periods of time, even in the most vulnerable infants. It uses multiple wavelengths of NIR light and relies on the distinct absorption spectra of oxygenated (O2Hb) and deoxygenated. NIRS offers the ability to assess target organ blood flow. It offers additional information regarding organ perfusion, which supplements data provided by echocardiography and other modalities. In preterm infants, NIRS-derived fractional tissue oxygen extraction and regional cerebral oxygen saturation reference values, particularly over the first 72 hours of life, are emerging. NIRS is being used in many centers including ours, in an ad-hoc manner. In a multicenter, randomized, controlled trial, infants monitored with NIRS and treated for evolving cerebral hypoxia had a lower cerebral hypoxic burden when compared with infants who were not treated based on NIRS findings. The long-term benefit of this approach has yet to be elucidated.

There have been attempts to combine the TNE and NIRS studies in preterm neonates to guide management, showing benefits including reduced inotrope use and length of stay. There is a clear need for a systematic evaluation of the hemodynamic state using a combination of TNE, NIRS and clinical assessment that will result in better clinical understanding of the physiology especially during the transitional period by the neonatal clinicians. The assessment of ELGAN hemodynamics without considering data regarding systemic flow, cardiac output and organ perfusion is incomplete and may result in unnecessary and potentially harmful management strategies.

Various scoring measures have been used in neonates and children to objectively categorize the cardiovascular support using inotrope use as a surrogate. Vasoactive inotrope score (VIS) which provides a numerical sum of inotrope doses used, has been used in preterm infants to quantify cardiovascular support in the perioperative period. A more comprehensive score - Vasoactive Ventilation Renal score (VVR) that incorporates ventilation support and renal function assessment has been used to evaluate children during the perioperative period. There are no neonatal studies using VVR scores in the transitional period after birth.

The hypothesis is having a detailed hemodynamic understanding using a multimodal assessment will result in less inotrope use in ELGAN as evidenced by lower VVR and VIS scores.

Objectives:

Primary Objective:

1. To determine whether a multimodal hemodynamic monitoring using combined TNE and cerebral NIRS can reduce inotrope use as evidenced by decreasingVasoactive-Ventilation-Renal(VVR) scores in ELGAN within the first one week of life
2. To investigate whether a multimodal hemodynamic monitoring using combined TNE and cerebral NIRS can reduce the VIS scores in the subset of ELGANS receiving inotropes in the first 72hours of life

Secondary Objective

To validate the use of VVR scores during the neonatal transition period in ELGAN population

Study design: Non-blinded Randomized Control Trial

Study site: This study will be conducted at the Stollery Children Hospital (RAH-Site NICU) NICU which is a 69-bed unit that specializes in the care of very premature infants. On an average, about 150 ELGAN less than 29 weeks are admitted per year to the RAH-Site NICU for specialized neonatal care.

Methodology: This will be a Non-blinded Randomized Control Trial.

The study will involve the following steps (APPENDIX 1)

1. The study population will be assigned by simple randomization to either Study arm to receive multimodal hemodynamic assessment using the study guideline (APPENDIX 5) or Standard arm to be treated according to the standard approach operative in the Neonatal Intensive Care Unit (NICU) of the Royal Alexandra Hospital.
2. ELGANs recruited into

A) Standard arm:

1. .Continuous cardiorespiratory monitoring using ECG leads or via an arterial line, and pulse oximetry and intermittent non-invasive blood pressure monitoring as standard of care in the NICU. Continuous arterial blood pressure monitoring will also be obtained as appropriate when an arterial line has been placed under the clinical team's discretion.
2. .TNE studies will be performed at the discretion of clinical team for concerns on cardiorespiratory status of the study population.
3. . Cerebral NIRS monitoring for regional Cerebral Oxygen saturation (rScO2) using Neonatal sensors attached to the forehead of the infant as per current practice
4. . The current treatment protocol for hemodynamic compromise at our NICU is starting inotropic support if Mean Blood Pressure is less than the gestational age of the infant in the first 72hours of life.

B) Study Arm:

1. ELGANs recruited to the study group will have the same monitoring outlined in 2a in a standardized manner. Zubrow's Normative BP chart will be used and MBP less than the third centile for the gestational age will be taken as low BP for the study
2. .Continuous cerebral NIRS monitoring for regional Cerebral Oxygen saturation (rScO2) using Neonatal sensor will be attached to the forehead of the infant (APPENDIX 2) for the first 72 hours of life.
3. .Hemodynamic assessment using TNE (APPENDIX 3) will be performed at 18-24 hours and 66-72 hours of life. Additional TNE studies will be performed at the discretion of clinical team for concerns on cardiorespiratory status of the study population.
4. .A hemodynamic report will be provided by the research team integrating the findings of the multimodal monitoring (ie Cardio-respiratory parameters, NIRS and TNE) within the clinical context (APPENDIX 5). No management suggestions will be provided in the report

   4.All neonates will have standardized assessment for lead related skin abrasions as per standard practice, neonatal pain and stress assessment (NPASS score) as part of their standard care

   5.Developmentally support care will be given by the support person during the TNE assessment as per standard unit practice

   6.The discontinuation of either or both NIRS and TNE will depend on the discretion of clinical team. Reason for the discontinuation will be sorted. This does not constitute a deviation from the study protocol.

   7.The admission, 24hrs, 48 hours, 72 hours and 7days mean and median VVR and VIS scores will be calculated in both Study and Standard arms. (APPENDIX 4)

   8.Urine output will be monitored during the study period as a surrogate for renal function and urine output less than 1ml/k/hr will be considered as oliguria.

   9.Score for Neonatal Acute Physiology with Perinatal Extension-II (SNAPPE-II) score which is a validated disease severity score in preterm babies will be calculated in both study and standard arm at admission, 72hours and 7days of life.

   10.Data on NIRS changes with normal saline bolus and blood products will also be collected in the study arm whenever appropriate.

   Data collection: The following patient demographics will be recorded: gestation, birth weight, type of pregnancy, type of delivery, antenatal morbidities (Pregnancy Induced Hypertension, placental abruption, chorio-amnionitis), antenatal steroids, antenatal Magnesium Sulphate, Apgar scores, and gender. Information will be collected about the active clinical issue and disease states at the time of the hemodynamic assessment. Data pertaining to cardiorespiratory support, ventilation requirement, inotropes requirement will be recorded during the first week of life. Data for the TNE cardiac function studies will be collected in a separate datasheet and continuous NIRS data will be collected for the first 72 hours of life. Major morbidity data like Chronic lung disease, Necrotizing Enterocolitis, Retinopathy of Prematurity, severe brain injury, Patent Ductus Arteriosus management and mortality will be collected for the purpose of validation of VVR score in the transitional neonatal period.

   Sample size:

   Sample size calculation for VVR scores

   Assuming 25% reduction in VVR in intervention arm with mean VVR score of 30 in control arm and 22.5 in intervention arm, sd-15; t test assuming sd1 = sd2 = sd; Ho: m2 = m1 versus Ha: m2 != m1

   Study parameters:

   alpha = 0.0500; power = 0.8000; delta = -7.5000; m1 = 30.0000; m2 = 22.5000

   sd = 15.0000

   Estimated sample sizes: N = 128; N per group = 64

   Sample size calculation for VIS scores

   Assuming 30% reduction in VIS in intervention arm with mean VIS score of 5 in control arm and 3.5 in intervention arm, sd-15; t test assuming sd1 = sd2 = sd; Ho: m2 = m1 versus Ha: m2 != m1

   Study parameters:

   alpha = 0.0500; power = 0.8000; m1 = 5 ; m2 = 3.5 sd = 15.0000

   Estimated sample sizes: N = 56; N per group = 28

   Analysis: All statistical analyses will be performed with the intercooled Stata Version 14.0 (College Station, Texas). All data will be anonymized for analysis. All the tests will be two-sided (where applicable) and significance will be defined as p-value <0.05. Univariate and bivariate analysis will be done to describe the sample. Categorical variables will be compared by Fisher's exact test and continuous variables by Student's t-test (two-sided). Logistic and linear regression models will be developed using statistical techniques to examine the association between arterial blood pressure, Cerebral oxygen saturation, the use of inotropes, VVR and VIS scores. Receiver Operating Curve will be used for the purpose of validation of the VVR scores in neonates during the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies less than 29 weeks (ELGAN)
* Babies born in Royal Alexandra Hospital(RAH) and admitted to RAH-NICU for first 7days of life

Exclusion Criteria:

* Structural heart diseases
* Major congenital disorder or chromosomal disorder

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Peak and Mean Vasoactive-Ventilation-Renal scores in both groups | at 7 days of life
  Higher the scores, higher the cardiovascular support
Peak and Mean Vasoactive Inotrope scores in both groups | at 7days of life
  Higher the scores, higher the cardiovascular support

SECONDARY OUTCOMES:
Duration of mechanical ventilation | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Total number of Days in the hospital | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Number of Participants with Chronic Lung Disease | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Number of Participants with Necrotizing Enterocolitis | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Number of Participants with Retinopathy Of Prematurity | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Number of Participants with severe brain injury | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Number of Participants with Patent Ductus Arterious | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period
Number of deaths | through study completion, an average of 44 weeks corrected gestation
  for the purpose of Validation of Vasoactive-Ventilation-Renal scores in the transition neonatal period

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Kumaran, Principal Investigator — University of Alberta; Po-Yin Cheung, Principal Investigator — University of Alberta; Matthew Hicks, Principal Investigator — University of Alberta; Abbas Hyderi, Principal Investigator — University of Alberta; Renjini Lalitha Kumari, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital-NICU, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lalitha R, Bitar E, Hicks M, Surak A, Hyderi A, Pepper D, Cheung PY, Kumaran K. Multimodal Monitoring of Hemodynamics in Neonates With Extremely Low Gestational Age: A Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e254101. doi: 10.1001/jamanetworkopen.2025.4101. PMID 40202760